CLINICAL TRIAL: NCT03193632
Title: The Novel Use of Point of Care Ultrasound to Predict Resting Energy Expenditure in Critically Ill Patients by Measuring Lean Body Mass Using Musculo-skeletal Ultrasound
Brief Title: Predicting Resting Energy Expenditure in Critically Ill Patients by Measuring Lean Body Mass by US
Status: Completed | Type: Observational
Sponsor: Eslam Ayman Mohamed Shawki (Other)
Responsible Party: Sponsor-Investigator, Eslam Ayman Mohamed Shawki, Lecturer of anesthesia, SICU & Pain Management, Cairo University
Organization: Cairo University (Other)
Other Study IDs: LBM_REE
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Resting Energy Expenditure
Keywords: lean body mass; resting energy expenditure; oxygen consumption; Indirect calorimetry; carbon dioxide excretion; respiratory quotient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Study group: critically-ill patients who will be admitted to the surgical ICU for ventilatory support and will be expected to continue for more than one day US Muscle layer thickness (MLT) estimation will be used to estimate LBM and REE estimation by indirect calorimetry will be performed
  Interventions: Diagnostic Test: US Muscle layer thickness (MLT) estimation; Diagnostic Test: REE estimation by indirect calorimetry

INTERVENTIONS:
Diagnostic Test: US Muscle layer thickness (MLT) estimation — Three measurements will be made at each of three sites; mid-upper arm, forearm and thigh anteriorly and the mean value will be calculated. Measurement sites will be marked with indelible ink to ensure day-to-day consistency.
  1. Thigh: MLT of the quadriceps femoris muscle (M. Vastus intermedius and M. rectus femoris) will be assessed bilaterally
  2. Mid-upper arm: Muscle layer thickness will be measured over the biceps,midway between the tip of the acromion and the tip of the olecranon
  3. Forearm: A point midway between the antecubital skin crease and the ulnar styloid was marked and muscle thickness down to the interosseus membrane
Diagnostic Test: REE estimation by indirect calorimetry — REE will be calculated using indirect calorimetry via metabolic module on General Electric ventilator (Engstrom Carestation and Carescape R860, GE Health care, USA) All indirect calorimetric measurements will be done using standardized technique. Gas calibration will be performed before each measurement, and the measurements will last for at least 30 minutes. Measurements will be taken with the patient lying supine and ventilator settings left unchanged for at least 60 minutes ahead of indirect calorimetry. The REE will be calculated during the first 24 hours of admission to ICU.

SUMMARY:
The study aims to correlate Lean Body Mass (LBM) Evaluated by Musculoskeletal Ultrasound with Resting Energy Expenditure (REE) measured by Indirect Calorimetry and to generate a predictive equation of REE based on LBM, in addition to identifying other factors that may affect REE such as age, gender, and severity scores.

DETAILED DESCRIPTION:
Caloric needs in critically-ill patients fluctuate significantly over the course of the disease which might expose patients to either malnutrition or overfeeding.Malnutrition is associated with deterioration of lean body mass (LBM), poor wound healing, increased risk of nosocomial infection, and weakened respiratory muscles. On the other hand overfeeding in medically compromised patients can promote lipogenesis, hyperglycemia, and exacerbation of respiratory failure. Many factors may affect the resting energy expenditure (REE) through manipulation of oxygen consumption (VO2). One of the strongest determinants of REE is the LBM.

A measurement of muscle mass and changes in muscle mass could thus provide an index of LBM in critically ill patients. At present, computerized tomography, magnetic resonance imaging and dual-energy X-ray absorptiometry (DXA) are widely used as reference methods for evaluating LBM in vivo. However, these methods are impractical in critically ill patients. More practically, ultrasound scanning is a simple, portable, safe, and a low-patient burden technique. Several studies found that the use of ultrasound can be a good estimate to LBM.

Indirect calorimetry remains the accepted standard for determining the REE in the critically ill. Indirect calorimetry measures oxygen consumption(VO2) and carbon dioxide excretion (VCO2 ) (both in mL/min), which are used to calculate the respiratory quotient and the resting energy expenditure. Although, the measured LBM has been shown as an important determinant of REE, there was no previous study tested the relationship between estimated LBM by ultrasound-based muscle thickness measurement and REE.

ELIGIBILITY:
Inclusion Criteria:

- Patient requiring ventilatory support > 24 hours

Exclusion Criteria:

* Patient who will require FIO2 more than 0.6.
* Air leak from the chest tube.
* Patient with body temperature > 39oC.
* Patients with known endocrine dysfunction.
* Patients on parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically-ill patients who will be admitted to the surgical ICU for ventilatory support and will be expected to continue more than one day
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
correlation between LBM derived from ultrasound MLT and REE by indirect calorimetry | 24 hours of ICU admission
  The correlation of the LBM derived from ultrasound MLT to the REE measured within 24 hours of ICU admission with indirect calorimetry

SECONDARY OUTCOMES:
Predictive equation for REE based on US measurement of MLT | 24 hours of ICU admission
  generation of predictive equation of REE based on ultrasound measurement of MLT
Estimation of the effect of severity scores on the REE | 24 hours of ICU admission
  Estimation of the effect of severity scores on the REE

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Cairo University teaching hospitals (Kasr Alainy), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rubinson L, Diette GB, Song X, Brower RG, Krishnan JA. Low caloric intake is associated with nosocomial bloodstream infections in patients in the medical intensive care unit. Crit Care Med. 2004 Feb;32(2):350-7. doi: 10.1097/01.CCM.0000089641.06306.68. PMID 14758147
- [Background] Covelli HD, Black JW, Olsen MS, Beekman JF. Respiratory failure precipitated by high carbohydrate loads. Ann Intern Med. 1981 Nov;95(5):579-81. doi: 10.7326/0003-4819-95-5-579. PMID 6794409
- [Background] Walker RN, Heuberger RA. Predictive equations for energy needs for the critically ill. Respir Care. 2009 Apr;54(4):509-21. PMID 19327188
- [Background] Fung EB. Estimating energy expenditure in critically ill adults and children. AACN Clin Issues. 2000 Nov;11(4):480-97. doi: 10.1097/00044067-200011000-00002. PMID 11288413
- [Background] Campbell IT, Watt T, Withers D, England R, Sukumar S, Keegan MA, Faragher B, Martin DF. Muscle thickness, measured with ultrasound, may be an indicator of lean tissue wasting in multiple organ failure in the presence of edema. Am J Clin Nutr. 1995 Sep;62(3):533-9. doi: 10.1093/ajcn/62.3.533. PMID 7661114
- [Background] Sanada K, Kearns CF, Midorikawa T, Abe T. Prediction and validation of total and regional skeletal muscle mass by ultrasound in Japanese adults. Eur J Appl Physiol. 2006 Jan;96(1):24-31. doi: 10.1007/s00421-005-0061-0. Epub 2005 Oct 19. PMID 16235068
- [Background] Pineau JC, Guihard-Costa AM, Bocquet M. Validation of ultrasound techniques applied to body fat measurement. A comparison between ultrasound techniques, air displacement plethysmography and bioelectrical impedance vs. dual-energy X-ray absorptiometry. Ann Nutr Metab. 2007;51(5):421-7. doi: 10.1159/000111161. Epub 2007 Nov 20. PMID 18025814
- [Background] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Background] Muller MJ, Illner K, Bosy-Westphal A, Brinkmann G, Heller M. Regional lean body mass and resting energy expenditure in non-obese adults. Eur J Nutr. 2001 Jun;40(3):93-7. doi: 10.1007/s003940170008. PMID 11697446